CLINICAL TRIAL: NCT04868526
Title: Dietary Intervention to Mitigate Adverse Consequences of Night Work
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Frank AJL Scheer, PhD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2021P000683; R01HL153969 (NIH)
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Dietary Habits
Keywords: Night shift work; Glucose tolerance
MeSH Terms: conditions — Feeding Behavior | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-Dietary Intervention (Experimental): Control condition first, then the Dietary intervention. Since this is a single blind study, the details of the dietary interventions cannot be released during recruitment stage but will be made public once enrollment closes.
  Interventions: Behavioral: dietary intervention
- Dietary intervention-Control (Experimental): Dietary intervention first, then the Control condition. Since this is a single blind study, the details of the dietary interventions cannot be released during recruitment stage but will be made public once enrollment closes.
  Interventions: Behavioral: dietary intervention

INTERVENTIONS:
Behavioral: dietary intervention — Research participants will be assigned to two dietary conditions.

SUMMARY:
The goal of this clinical trial is to test whether our dietary intervention can prevent or lessen the negative health effects of night shift work in healthy participants.

Participants will:

* complete 2 inpatient stays
* be provided with identical meals
* have frequent blood draws
* provide urine, saliva, stool and rectal swab samples

DETAILED DESCRIPTION:
Shift work increases the risk for diabetes possibly due to the adverse metabolic effects of circadian misalignment. As shift work is not foreseen to disappear, the development of individually-targeted therapies for metabolic health in these vulnerable shift workers is urgently needed. This research will determine whether our dietary intervention can mitigate the adverse metabolic effects of circadian misalignment, which may help in the design of evidence-based dietary interventions to improve the metabolic health in shift workers.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 yr old
* BMI 20.0-29.9
* European/Hispanic/African-American ancestry
* No acute, chronic or debilitating medical conditions (e.g. metabolic, cardiovascular, respiratory, neurological, cancers, etc.)

Exclusion Criteria:

* Currently smoking/vaping or 5 or more years of smoking/vaping
* History of drug or alcohol dependency
* History of psychiatric illness or disorder

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in glucose tolerance from Baseline to Test Day | Baseline (Day 2) and Test Day (Day 4)
  Change in incremental glucose area under the curve (AUC) from a mixed meal test.
Changes in microbial community structure/composition/function of oral and gut microbiome from Baseline to Test Day | Baseline (Day 2) and Test Day (Day 4)
  Shotgun metagenomics sequencing or 16S rRNA sequencing of saliva, stool, and rectal swab samples will provide in-depth interrogation of the microbial community structure, composition, and function.

SECONDARY OUTCOMES:
Change in insulin sensitivity (Oral Minimal Model method) from Baseline to Test Day | Baseline (Day 2) and Test Day (Day 4)
  Oral Minimal Model method estimates insulin sensitivity based on blood glucose and insulin levels from a mixed meal test.
Change in levels of serum markers of gut microbiota from Baseline to Test Day | Baseline (Day 2) and Test Day (Day 4)
  Levels of markers of gut microbiota (e.g. short chain fatty acids) will be measured in serum samples taken 3-hourly over 24 hr.
Change in levels of serum markers of intestinal barrier integrity from Baseline to Test Day | Baseline (Day 2) and Test Day (Day 4)
  Levels of markers of intestinal barrier integrity (e.g. zonulin, LPS, LBP) will be measured in serum samples taken 3-hourly over 24 hr.
Change in level of serum markers of inflammatory state from Baseline to Test Day | Baseline (Day 2) and Test Day (Day 4)
  Levels of markers of inflammatory state (e.g., cytokines) will be measured in serum samples taken 3-hourly over 24 hr.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Scheer, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No